CLINICAL TRIAL: NCT03223259
Title: Educating the Educator to Reduce Risk of Dance Student Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-00723
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Injuries
Keywords: Dance Injuries; Injury Prevention Workshops; Motor Skill Theory; Gross Motor Skills
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injury Prevention Workshops (Other): Subjects will attend two Injury Prevention Workshops
  Interventions: Behavioral: Injury Prevention Workshops

INTERVENTIONS:
Behavioral: Injury Prevention Workshops — Each workshop will last 90 minutes and consist of approximately 20-30 minutes of lecture, 30 minutes of movement, no more than 20 minutes for a pre-test (workshop 1) or post-test (workshop 2), and remaining time for Q&A.

SUMMARY:
A group of dance educators will attend two dance injury prevention workshops hosted by the Harkness Center for Dance Injuries (HCDI), NYU Langone Medical Center, during which participants will learn strategies to help them train their students in safe ways and impart injury prevention information through their dance classes to their students. The educators will take pre- and post-workshop tests to assess knowledge and perceptions of dance medicine. Several weeks later, participants will take a follow-up survey to assess knowledge implementation and workshop effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Teach dance to children in at least one private dance school
* Must be able to receive email and complete a survey online
* Must believe that students lack access to dance injury prevention resources
* Must teach at least one group of students that takes class from them a minimum of twice a week and must teach those students regularly in September and October, 2017.

Exclusion Criteria:

* Under the Age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Score on Injury Prevention Workshop Pre-Test and Post-Test | 20 Minutes
  The test will ask subjects questions about their dance teaching background and ascertain their current knowledge of dance anatomy and injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Rose, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States